CLINICAL TRIAL: NCT02995941
Title: Shoulder Symptom Irritability: A Single-Blinded Observational Study of Reliability and Construct Validity
Brief Title: Shoulder Symptom Irritability Scale: A Single-Blinded Observational Study
Acronym: SSIS
Status: Completed | Type: Observational
Sponsor: St. Luke's Hospital and Health Network, Pennsylvania (Other)
Collaborators: Arcadia University (Other); Nova Southeastern University (Other)
Responsible Party: Principal Investigator, Stephen Kareha, DPT, Director, Orthopaedic Physical Therapy Residency, St. Luke's Hospital and Health Network, Pennsylvania
Other Study IDs: 2016-61
Record Dates: First submitted 2016-12-10; First posted 2016-12-19 (Estimated); Last update posted 2019-09-20 (Actual); Status verified 2019-09

CONDITIONS: Shoulder Pain; Pain
Keywords: reliability; validity; classification; irritability; symptom; intensity; intervention
MeSH Terms: conditions — Shoulder Pain; Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Raters: No interventions will be administered. Raters will be state licensed as physical therapists working as outpatient physical therapists in the St. Luke's University Health Network.
- Patients: No interventions will be administered as a component of this study. Patients will be recruited from a convenience sample of consecutive patients presenting for physical therapy consultation for shoulder pain.

SUMMARY:
The purpose of this study is to examine the reliability and use of the shoulder symptom irritability classification system for the purposes of determining an appropriate treatment intensity to better help people with shoulder pain.

DETAILED DESCRIPTION:
Background Physical therapists regularly make decisions regarding intervention intensity based upon pathoanatomy, symptom irritability, and impairment identification, but the reliability and validity of classifying patients by symptom irritability is unknown.

Purpose Examine the reliability and use of the shoulder symptom irritability classification system for the purposes of determining an appropriate treatment intensity.

Design Prospective repeated-measures single-blinded design to determine reliability and a cross-sectional design will be utilized to aid in determining construct validity.

Methods Twenty-five (25) raters will be trained to make paired ratings in 90 subjects with primary complaints of shoulder pain. Raters will record the shoulder symptom irritability level and also select the appropriate intervention intensities for the subjects. Raters will also be asked to choose anticipated interventions for subjects.

Data Analysis Prevalence-adjusted, bias-adjusted Kappa for ordinal scales (PABAK-OS) will be the primary measure of reliability. Dependent upon the distribution of the data, other forms of Kappa may be utilized to analyze the data most appropriately. To determine differences in reliability between groups with and without clinical specialization, an independent t test will be utilized with α = 0.05. Lastly, analysis of variance with post-hoc analysis will be used to compare functional disability across different levels of irritability.

Significance This study addresses key gaps in the understanding of symptom irritability and how it relates to clinical decision making. It is expected that symptom irritability should logically drive intervention selection and intensity of rehabilitation interventions.

ELIGIBILITY:
Rater Group

Inclusion Criteria:

* State licensure as a physical therapist and regular clinical practice with patients with shoulder disorders, defined as a minimum of 500 clinical hours per year in an orthopaedic setting with >10% of patients with shoulder disorders

Exclusion Criteria:

* not meeting inclusion criteria

Patient Group

Inclusion Criteria:

* Presenting with a chief complaint of shoulder pain, not extending to the neck, for outpatient physical therapy consultation

Exclusion Criteria:

* Illiteracy in English and age less than 18 years. Additionally, subjects will be excluded from the study if they present with pain or symptoms distal to elbow, have had shoulder surgery on the symptomatic side in the past year, if active or passive cervical spine ROM reproduces shoulder pain, have a positive Spurling's test, or if they are unable to complete the patient reported functional questionnaires

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Raters will be recruited from outpatient physical therapists in the St. Luke's University Health Network.
  Patient subjects will be recruited from a convenience sample of consecutive patients presenting for physical therapy consultation for shoulder pain.
Sampling Method: Non-Probability Sample
Enrollment: 138 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Reliability of Shoulder Symptom Irritability Scale | Day 1 of data collection for each subject
  Two different raters will individually rate the shoulder symptom irritability of each patient. Raters will be blinded to the other's rating.

SECONDARY OUTCOMES:
Focus On Therapeutic Outcomes (FOTO) Functional Score | Day 1 of data collection for each subject
  The FOTO functional scale for shoulder disorders27 has a standard error of the mean (SEM) of 1. with a minimal detectable change with 95% confidence (MDC95) of 3.60-10.88 functional score units.
Penn Shoulder Score (PSS) | Day 1 of data collection for each subject
  The Penn Shoulder Score (PSS)has demonstrated good test-retest reliability (ICC2,1 = 0.94) with a SEM90 of 8.5. The MDC90 is 12.1, and the minimal clinically important difference (MCID) was found to be 11.4.
American Shoulder and Elbow Surgeons (ASES) Shoulder Score | Day 1 of data collection for each subject
  The ASES Shoulder Score has demonstrated good to excellent test-retest reliability (ICC = 0.61-0.96) with an SEM of 6.7. The MDC95 is 11.2,32 and the MCID was found to be 12.0.
Numeric Pain Rating scale | Day 1 of data collection for each subject
  The Numeric Pain Rating Scale (NPRS) has demonstrated good reliability (ICC2,1=0.74)and responsiveness (MDC = 2.5, MCID = 1.1) in subjects with shoulder pain34 and excellent reliability in an upper extremity orthopaedic population.
Intervention intensity | Day 1 of data collection for each subject
  This project will analyze intervention choices from the primary raters for each of the 90 subjects utilizing PABAK-OS for correlation and independent t-test for group differences. It is expected that those subjects with high irritability will be prescribed interventions aimed at minimizing the physical stress to the affected tissue(s), while those subjects with low irritability will be prescribed interventions at a higher intensity to address the physical impairments.

CONTACTS AND LOCATIONS:
Overall Officials: Alicia Fernandez-Fernandez, DPT, PhD, Study Chair — Nova Southeastern University; Stephen M Kareha, DPT, Principal Investigator — St. Luke's Hospital and Health Network, Pennsylvania
Locations (17):
- United States (17):
  - Physical Therapy at St. Luke's - Washington, Washington, New Jersey
  - Physical Therapy at St. Luke's - Hamilton, Allentown, Pennsylvania
  - Physical Therapy at St. Luke's - West End Medical Center, Allentown, Pennsylvania
  - Physical Therapy at St. Luke's - Bath, Bath, Pennsylvania
  - Physical Therapy at St. Luke's - St. Luke's North, Bethlehem, Pennsylvania
  - Physical Therapy at St. Luke's - Sports Medicine and Rehab Center, Bethlehem, Pennsylvania
  - Physical Therapy at St. Luke's - Center Valley, Center Valley, Pennsylvania
  - Physical Therapy at St. Luke's - Forks, Easton, Pennsylvania
  - Physical Therapy at St. Luke's - Anderson, Easton, Pennsylvania
  - Physical Therapy at St. Luke's - Emmaus, Emmaus, Pennsylvania
  - Physical Therapy at St. Luke's - Hellertown, Hellertown, Pennsylvania
  - Physical Therapy at St. Luke's - Macungie, Macungie, Pennsylvania
  - Physical Therapy at St. Luke's - Northampton, Northampton, Pennsylvania
  - Physical Therapy at St. Luke's - Orefield, Orefield, Pennsylvania
  - Physical Therapy at St. Luke's - Quakertown, Quakertown, Pennsylvania
  - Physical Therapy at St. Luke's - Stroudsburg, Stroudsburg, Pennsylvania
  - Physical Therapy at St. Luke's - Wind Gap, Wind Gap, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kareha SM, McClure PW, Fernandez-Fernandez A. Reliability and Concurrent Validity of Shoulder Tissue Irritability Classification. Phys Ther. 2021 Mar 3;101(3):pzab022. doi: 10.1093/ptj/pzab022. PMID 33481995
- See also: Shoulder Symptom Irritability Scale Rater Training — https://youtu.be/a-QiJ5-bKKQ

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2016-10-31): https://cdn.clinicaltrials.gov/large-docs/41/NCT02995941/Prot_SAP_ICF_000.pdf